CLINICAL TRIAL: NCT02385045
Title: i-Scan for the Detection of Helicobacter Pylori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14SM2185
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narrow band imaging (Placebo Comparator): Narrow band imaging function (Olympus endoscopes)
  Interventions: Device: narrow band imaging
- i-scan imaging (Experimental): i-scan imaging (Pentax endoscopes)
  Interventions: Device: i-scan

INTERVENTIONS:
Device: i-scan — i-scan function is located on the head of the Pentax endoscopes
  Arms: i-scan imaging
Device: narrow band imaging — narrow band imaging function is located on the head of Olympus endoscopes
  Arms: Narrow band imaging

SUMMARY:
This study aims to assess whether iScan, an intra-endoscopic imaging technique is an accurate and reliable tool in detecting and characterising Helicobacter pylori (H pylori) and comparing this to standard endoscopic imaging with white light endoscopy (WLE), narrow band imaging (NBI) and histology.

DETAILED DESCRIPTION:
The ultimate goal of endoscopy will be the 'optical biopsy' i.e. forgoing the need to take histological samples to make a diagnosis in order to reduce complication rates, cost and time. There are a number of imaging techniques which promise to improve our diagnostic rates for pathology, but there have been few comparative studies.

This is randomized controlled parallel trial in a 1:1 ratio with examination of the upper gastrointestinal tract with WLE followed by either NBI or iscan.

(Note: Prior to commencement of the study, technical issues and operational changes in our organisation forced the removal of the Pentax 'i-scan' endoscopes. Recruitment to this arm was anticipated, but was ultimately not possible.)

Patients attending the department for routine examinations for dyspepsia and abdominal pain will be randomised into 2 study arms (1WLE and NBI, and the other - WLE and iscan).

The investigator carrying out the procedure will be blinded to the indication for the procedure until a full examination with both white light endoscopy and either NBI or iscan has been used as this could lead to bias. They will determine if H pylori is present, and if so the severity of infection with WLE and again with either NBI or iscan depending on their study arm. Histopathological confirmation of H pylori and an assessment to the degree of infection will be assessed with samples taken using the updated Sydney system (5 gastric samples from different parts of the stomach).

The endoscopists reviewing the images will be blinded to all patient information and indications throughout the study period. Questionnaires will then be given to the endoscopists to determine what endoscopic features led them to their diagnosis.

ELIGIBILITY:
Inclusion Criteria:

• All patients attending for a routine diagnostic endoscopic procedure at St Mary's Hospital NHS Trust for dyspepsia and abdominal pain

Exclusion Criteria:

* Patients attending for a therapeutic endoscopic procedure e.g. variceal banding, stent insertion, balloon dilatation.
* Patients with a known diagnosis e.g. upper gastrointestinal cancer
* Patients previously treated with HP eradication therapy
* Patients who had taken PPI, H2 receptor antagonists and antibiotics within 4 weeks
* Patients with acute gastrointestinal bleeding
* Patients who'd had previous gastric surgery
* Patients with chronic liver disease
* Patients with abnormal coagulation or any other contra-indication to use of standard biopsy in routine diagnostic endoscopic procedures
* Patients who are unable or unwilling to give informed consent
* Patients under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Teare, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Glover B, Teare J, Patel N. Assessment of Helicobacter pylori status by examination of gastric mucosal patterns: diagnostic accuracy of white-light endoscopy and narrow-band imaging. BMJ Open Gastroenterol. 2021 Aug;8(1):e000608. doi: 10.1136/bmjgast-2021-000608. PMID 34353822

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Narrow Band Imaging
Started | 157
Completed | 153 (4 patients could not complete endoscopy as planned)
Not Completed | 4
Not completed — Endoscopy could not be completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Narrow Band Imaging
Number analyzed (Participants) | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 106
  >=65 years | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 66
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 153

OUTCOME MEASURES:

1. Primary Outcome: Successful Diagnosis of Helicobacter Pylori Using Imaging Modality
Description: The endoscopic assessment of the presence of H pylori using standard endoscopy plus NBI will be compared to histological assessment. Inter-observer variability of assessment of the presence of H pylori will be compared between endoscopic imaging techniques
Time Frame: 1 year
Population: All patients presenting for endoscopy who were recruited to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Band Imaging
Number analyzed (Participants) | 153
Participants
  H Pylori Positive | 28
  H Pylori Negative | 125

ADVERSE EVENTS:
Time Frame: 1 year
Description: Patients developing adverse events were to be identified either at the time of endoscopy, or on review of patient records at the time of study reporting.
Arm/Group | Narrow Band Imaging
All-Cause Mortality (participants affected / at risk) | 0/153
Serious Adverse Events (participants affected / at risk) | 0/153
Other Adverse Events (participants affected / at risk) | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes